CLINICAL TRIAL: NCT07201402
Title: Prospective Long-term Study of Etonogestrel Contraceptive Implant Insertion at an Alternative Scapular Site
Brief Title: Long Term Evaluation of Scapular-inserted Contraceptive Implants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Aaron Lazorwitz, Associate Professor of Obstetrics, Gynecology and Reproductive Sciences, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000040944; R56HD117869 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Contraception
Keywords: contraceptive implant; scapular insertion site; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Reproductive age females (Experimental): All study participants will be reproductive age females interested in using an etonogestrel contraceptive implant
  Interventions: Drug: Scapular-site insertion of etonogestrel contraceptive implant

INTERVENTIONS:
Drug: Scapular-site insertion of etonogestrel contraceptive implant — Participants will undergo insertion of the etonogestrel contraceptive implant subdermally over the inferior edge of their non-dominant scapula

SUMMARY:
This study aims to evaluate long-term outcomes when the etonogestrel contraceptive implant is inserted at an alternative site located over the scapular. The study will evaluate the pharmacokinetics (i.e., drug levels) and side effect profiles of participants who have an etonogestrel contraceptive implant inserted at this alternative scapular site over the course of at least two years.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Sex assigned at birth must be Female
4. Aged 18-45 years
5. In good general health as evidenced by medical history and no need for regular intensive medical interventions (e.g., inpatient admissions, surgical treatments). The Principal Investigator will be responsible for determining good general health for potential participants with complicated medical histories
6. Interest and willingness to use an etonogestrel contraceptive implant
7. Negative pregnancy test at the time of study enrollment and not planning to become pregnant in the next 36 months
8. Willing to abstain from medications and supplements known to induce/inhibit CYP3A (e.g., rifampin, carbamazepine, ketoconazole, St. John's wort) during the study. In the inducer/inhibitor CYP3A medication is a prescribed medication, individuals must provide the prescriber information for the PI to confirm it is safe for this medication to be abstained during the study
9. Body-mass index ≥18.5kg/m2

Exclusion Criteria:

1. Contradictions to the use of the ENG implant based on the CDC Medical Eligibility Criteria guidelines for any conditions with a category 3 or 4 recommendation

   1. Current breast cancer or personal history of breast cancer
   2. Malignant liver tumor (hepatocellular carcinoma)
2. Known liver conditions that could affect drug metabolism (e.g., cirrhosis, hepatitis)
3. Currently taking and unable or unwilling to abstain from any medications or supplements known to be CYP3A inducers/inhibitors
4. Current use of a progestin-only contraceptive method containing desogestrel or etonogestrel

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Serum etonogestrel concentrations | Every 6 months after insertion of the etonogestrel implant for up to 36 months (3 years)
  Serum etonogestrel concentrations measured using a validated LC-MS assay

SECONDARY OUTCOMES:
Progestin-related side effects | Every 6 months after insertion of the etonogestrel contraceptive implant for up to 36 months (3 years)
  Assessment of common progestin-related side effects (e.g., nausea, headaches, bloating) using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lazorwitz, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Serum etonogestrel concentrations and progestin-related side effect outcomes will be shared using NICHD DASH at the conclusion of the study
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP will be uploaded to clinicaltrials.gov within one year of completion of all study procedures and made available indefinitely
Access Criteria: Access to IPD uploaded to NICHD DASH will be handled via the existing DASH access protocols
URL: https://dash.nichd.nih.gov

REFERENCES:
- [Background] Clure C, Sheeder J, Lazorwitz A. Pilot study of a novel, alternative subdermal scapular insertion site for the etonogestrel contraceptive implant. Contraception. 2024 Jul;135:110442. doi: 10.1016/j.contraception.2024.110442. Epub 2024 Mar 27. PMID 38552822